CLINICAL TRIAL: NCT02534350
Title: A Phase 2b, Randomized, Controlled Trial Evaluating GS-5806 in Lung Transplant (LT) Recipients With Respiratory Syncytial Virus (RSV) Infection
Brief Title: Presatovir in Lung Transplant (LT) Recipients With Respiratory Syncytial Virus (RSV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-218-1797; 2015-002287-16 (EudraCT Number)
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Respiratory Syncytial Virus (RSV); Antiviral; Lung Transplant
MeSH Terms: interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Presatovir (Experimental): Presatovir 200 mg (4 x 50 mg) on Day 1, followed by 100 mg (2 x 50 mg) from Day 2 to Day 14
  Interventions: Drug: Presatovir
- Placebo (Placebo Comparator): Placebo tablets for a total of 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Presatovir — Tablets administered orally or via nasogastric (NG) tube once daily
  Other Names: GS-5806
  Arms: Presatovir
Drug: Placebo — Tablets administered orally or via NG tube once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of presatovir on nasal respiratory syncytial virus (RSV) viral load in RSV-positive lung transplant (LT) recipients with acute respiratory symptoms.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females ≥18 years of age who have received a LT (single or double) or heart/lung transplant > 90 days prior to Screening
* Confirmed to be RSV-positive by local polymerase chain reaction (PCR) testing (starting from when the upper or lower respiratory tract sample is obtained) ≤ 7 days prior to investigational medicinal product (IMP) administration on Day 1/Baseline
* New onset or acute worsening, if the symptom is chronic, of at least 1 of the following respiratory symptoms ≤ 7 days prior to IMP administration on Day 1/Baseline: nasal congestion, earache, runny nose, cough, sore throat, shortness of breath, or wheezing
* A negative local urine or serum pregnancy test for female subjects of childbearing potential at Screening, within 1 day prior to IMP administration. When available, existing local pregnancy test results obtained prior to Screening may be used, provided the testing was completed within 1 day prior to IMP administration
* Agreement from male and female subjects of childbearing potential who engage in heterosexual intercourse to use protocol specified method(s) of contraception

Key Exclusion Criteria:

Related to concomitant or previous medication use:

* Use of any non-marketed (according to region) investigational agents within 30 days, OR use of any investigational monoclonal anti-RSV antibodies within 4 months or 5 half-lives of Screening, whichever is longer, OR use of any prior investigational RSV vaccines
* Use of a strong or moderate cytochrome P450 enzyme (CYP) inducer including but not limited to rifampin, St. John's Wort, carbamazepine, phenytoin, efavirenz, bosentan, etravirine, modafinil, and nafcillin, within 2 weeks prior to the first dose of IMP

Related to transplant history:

• Recipient of any other organ transplant prior to Screening, with the exception of a LT (single or double) or heart/lung transplant

Related to medical condition at Screening:

* Known viral coinfection (including but not limited to influenza, metapneumovirus, human rhinovirus, parainfluenza, cytomegalovirus, or coronavirus) in the upper or lower respiratory tract ≤ 14 days prior to Screening unless discussed with the medical monitor and deemed acceptable
* Active systemic infection or infectious pneumonia of any etiology (ie, bacterial, viral [other than RSV] or fungal), including aspiration pneumonia, that is considered clinically significant by the investigator unless discussed with the medical monitor and deemed acceptable

Related to laboratory values:

* Clinically significant kidney dysfunction as defined by: An estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease (MDRD) study 4 parameter equation obtained from screening laboratory measurements or via local laboratory measurements obtained ≤ 7 days prior to Screening. The eGFR may be manually calculated or the reported eGFR value may be used, but any automatically calculated eGFR must be calculated using the MDRD equation.
* Clinically significant liver function test abnormalities as defined by an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) obtained in screening laboratory measurements or via local laboratory measurements obtained ≤ 7 days prior to Screening
* Clinically significant elevations in total bilirubin (TB), as determined by the investigator

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (28):
- United States (17):
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Stanford, California
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Seattle, Washington
- Australia (3):
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Murdoch, Western Australia
- Belgium (2):
  - Brussels
  - Yvoir
- Toronto, Ontario, Canada
- Strasbourg, France
- Germany (2):
  - Hanover
  - Munich
- Rotterdam, Netherlands
- Cambridge, United Kingdom

REFERENCES:
- [Derived] Gottlieb J, Torres F, Haddad T, Dhillon G, Dilling DF, Knoop C, Rampolla R, Walia R, Ahya V, Kessler R, Budev M, Neurohr C, Glanville AR, Jordan R, Porter D, McKevitt M, German P, Guo Y, Chien JW, Watkins TR, Zamora MR. A randomized controlled trial of presatovir for respiratory syncytial virus after lung transplant. J Heart Lung Transplant. 2023 Jul;42(7):908-916. doi: 10.1016/j.healun.2023.01.013. Epub 2023 Feb 7. PMID 36964084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at sites in Europe, North America, and Australia.The first participant was screened on 31 December 2015 and the last study visit occurred on 27 September 2017.
Pre-assignment Details: 111 participants were screened.
Groups:
- Presatovir: 200 mg (4 x 50 mg) on Day1/Baseline followed by 100 mg (2 x 50 mg) on Days 2 through 14 administered orally or via nasogastric (NG) tube once daily
- Placebo: Tablets administered orally or via NG tube once daily for 14 days
Period: Overall Study
Arm/Group | Presatovir | Placebo
Started | 41 | 20
Completed | 37 | 20
Not Completed | 4 | 0
Not completed — Randomized But Not Treated | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrew Consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 full dose of study drug
Groups:
- Presatovir: 200 mg (4 x 50 mg) on Day1/Baseline followed by 100 mg (2 x 50 mg) on Days 2 through 14 administered orally or via NG tube once daily
- Total: Total of all reporting groups
Arm/Group | Presatovir | Placebo | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.54) | 55.1 (14.23) | 56.0 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 21 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 36 | 19 | 55
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 36 | 16 | 52
  Other | 1 | 1 | 2
  Not Permitted | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 1
  Netherlands | 1 | 0 | 1
  Belgium | 2 | 2 | 4
  United States | 25 | 12 | 37
  United Kingdom | 1 | 0 | 1
  Australia | 2 | 1 | 3
  France | 2 | 0 | 2
  Germany | 7 | 4 | 11
Nasal Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  log10 copies/mL
    number analyzed (Participants) | 37 | 20 | 57
    (all) | 5.88 (2.088) | 6.59 (2.092) | 6.13 (2.098)
inFLUenza Patient-Reported Outcome (FLU-PRO) Score [Mean (Standard Deviation); unit: units on a scale] — Flu-PRO Score was calculated as the mean of 38 individual scores. Individual scores ranged from 0 (no symptoms) to 4 (worst symptoms) for the 5-point severity scale and 0 (never) to 4 or more times (always) for the 5-point frequency scale. Population: Participants in the Safety Analysis Set with available data were analyzed.
  units on a scale
    number analyzed (Participants) | 37 | 18 | 55
    (all) | 2.05 (0.607) | 2.11 (0.684) | 2.07 (0.628)
The Forced Expiratory Volume in One Second (FEV1) % Predicted [Mean (Standard Deviation); unit: percent FEV1] — Population: Participants in the Safety Analysis Set with available data were analyzed.
  percent FEV1
    number analyzed (Participants) | 40 | 19 | 59
    (all) | 63.64 (24.787) | 61.95 (18.625) | 63.10 (22.834)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Change in Viral Load From Day 1/Baseline Through Day 7 in Participants in the Full Analysis Set
Time Frame: Up to 7 days
Population: Participants in the Full Analysis Set (participants who received at least 1 full dose of study drug and had an RSV viral load ≥ lower limit of quantification (LLOQ) of the real-time quantitative polymerase chain reaction (RT-qPCR) assay in the Day 1 nasal sample, as determined by RT-qPCR at the central lab) with available data were analyzed .
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 35 | 19
log10 copies/mL | -0.73 (0.938) | -0.90 (0.815)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.72, ANCOVA; Treatment Difference = 0.10, 95% CI 2-sided [-0.43 to 0.63]

2. Primary Outcome: Time-Weighted Average Change in Viral Load From Day 1/Baseline Through Day 7 in a Subset of Participants in the Full Analysis Set Whose Duration of RSV Symptoms Prior to the First Dose of Study Drug is ≤ Median
Time Frame: Up to 7 days
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 16 | 11
log10 copies/mL | -0.83 (1.013) | -0.83 (0.757)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.76, ANCOVA; Treatment Difference = -0.12, 95% CI 2-sided [-0.94 to 0.69]

3. Secondary Outcome: Time-Weighted Average Change in FLU-PRO Score From Day 1/Baseline Through Day 7
Description: The Flu-PRO is a patient-reported outcome questionnaire utilized as a standardized method for evaluating symptoms of influenza. Flu-PRO Score was calculated as the mean of 38 individual scores. Individual scores ranged from 0 (no symptoms) to 4 (worst symptoms) for the 5-point severity scale and 0 (never) to 4 or more times (always) for the 5-point frequency scale. The mean values presented were calculated using the ANCOVA model and are adjusted for baseline value and stratification factor.
Time Frame: Up to 7 days
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 33 | 17
units on a scale | -0.27 (0.313) | -0.31 (0.298)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.86, ANCOVA; Treatment Difference = 0.01, 95% CI 2-sided [-0.12 to 0.15]

4. Secondary Outcome: Percent Change From Study Baseline in FEV1% Predicted Value
Description: FEV1 is defined as forced expiratory volume in the first second.
Time Frame: Baseline; Day 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 30 | 17
percent change | 22.69 (27.437) | 26.36 (23.312)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.60, ANCOVA; Treatment Difference = -3.25, 95% CI 2-sided [-15.58 to 9.08]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: Safety Analysis Set
Arm/Group | Presatovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/40 | 4/20
Other Adverse Events (participants affected / at risk) | 24/40 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=40) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=40) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Flatulence (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Fatigue (General disorders) | 4 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Nasal herpes (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 2
Chest X-ray abnormal (Investigations) | 0 | 1
Forced expiratory flow decreased (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 5 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2015-06-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT02534350/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02534350/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT02534350/SAP_002.pdf
  • Study Protocol: Amendment 2 (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT02534350/Prot_003.pdf